CLINICAL TRIAL: NCT00220961
Title: Actos Now for Prevention of Diabetes (ACT NOW)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: University of Texas (Other); Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Ralph DeFronzo, MD, Professor of Medicine, Chief of Diabetes, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 02-062A
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-06

CONDITIONS: Impaired Glucose Tolerance; Type 2 Diabetes
Keywords: Impaired Glucose Tolerance; Type 2 Diabetes; Prevention; Pioglitazone
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet similar to pioglitazone tablet
  Interventions: Drug: Placebo
- Pioglitazone (Active Comparator): Pioglitazone tablet similar to placebo tablet
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone tablets - 45 mg/day
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — Placebo tablets similar to pioglitazone tablets - 1 tablet/day
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether pioglitazone versus placebo can reduce the conversion rate of impaired glucose tolerance (IGT) to type 2 diabetes mellitus

DETAILED DESCRIPTION:
IGT is a prediabetic state. If IGT can be prevented from progressing to overt diabetes, the hyperglycemia-related complications of this devastating disease can be prevented. Subjects with IGT will be identified with an oral glucose tolerance test (OGTT). Eligible subjects also will have a measurement of first phase insulin secretion and insulin sensitivity using the frequently sampled intravenous glucose tolerance test (FSIVGTT) and carotid intimal media thickness using carotid ultrasound. Following these measurements subjects will be randomized to receive pioglitazone or placebo and they will return every 3 months for determination of fasting plasma glucose (FPG) concentration and interim medical history. Recruitment will take place over 15 months. From the time that the recruitment period ends, subjects will be followed for a total of 24 months on pioglitazone or placebo. The OGTT will be repeated at 15,27, and 39 months, or if the FPG is ≥ 126 mg/dl on the 3-month follow up visits. If the diagnosis of diabetes is established before month 39 or at month 39, the FSIVGTT and carotid ultrasound will be repeated. At 39 months, subjects will be washed out of pioglitazone or placebo and the OGTT, FSIVGTT, and carotid ultrasound will be repeated at month 45.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* All ethnic groups
* 18 years of age and older
* Impaired glucose tolerance by glucose tolerance test (fasting glucose 95-125 mg/dl and 2 hr glucose of 140-199 mg/dl)
* At least one of the following:

  * One or more components of the insulin resistance syndrome (HDL < 40 mg/dl in females and <35 mg/dl in males, fasting triglycerides > 150 mg/dl, blood pressure > 135/85 mmHg, BMI > 24 kg/m2, waist circumference > 102 cm in men and > 88 cm in women)
  * One or more first degree relatives with type 2 diabetes
  * History of gestational diabetes
  * Polycystic ovarian disease
  * Minority ethnic background (Mexican American, African American, Asian and Pacific Islanders, Native American)

Exclusion Criteria:

* Type 2 diabetes
* Previously treated with thiazolidinediones (ever) or metformin (within one year)
* Previously treated with a sulfonylurea, a meglitinide, an alpha glucosidase inhibitor for more than a week within last year or within the 3 months prior to randomization
* Previously treated with insulin (other than during pregnancy) for more than one week within the last year or within the 3 months prior to randomization
* Cardiovascular disease
* Hospitalization for treatment of heart disease or stroke in past 6 months
* New York Heart Association Functional Class > 2
* Left bundle branch block or third degree AV block
* Aortic stenosis
* SBP > 180 mmHg or DBP > 105 mmHg
* Renal disease
* Anemia
* Hepatitis
* GI diseases (pancreatitis, inflammatory bowel disease)
* Recent or significant abdominal surgery
* Advanced pulmonary disease
* Chronic infections
* Weight loss > 10% in past 6 months
* Pregnancy and childbearing
* Major psychiatric disorders
* Excessive alcohol intake
* Thiazide use > 25 mg per day
* Non-selective beta blockers
* Niacin
* Systemic glucocorticoids
* Weight loss or weight gain medication
* Thyroid disease-suboptimally treated
* Active endocrine diseases (Cushing's, acromegaly)
* Plasma triglycerides over 400 mg/dl (despite treatment)
* History bladder cancer
* Hematuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2004-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A. DeFronzo, M.D., Principal Investigator — Texas Diabetes Institute
Locations (8):
- United States (8):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - USC-Keck School of Medicine, Los Angeles, California
  - University of California San Diego-San Diego VA Medical Center, San Diego, California
  - Georgetown University, Washington D.C., District of Columbia
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - SUNY Health Science Center, Brooklyn, New York
  - University of Tennessee, Memphis, Tennessee
  - Texas Diabetes Institute, San Antonio, Texas

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751
- [Derived] Tripathy D, Schwenke DC, Banerji M, Bray GA, Buchanan TA, Clement SC, Henry RR, Kitabchi AE, Mudaliar S, Ratner RE, Stentz FB, Musi N, Reaven PD, DeFronzo RA. Diabetes Incidence and Glucose Tolerance after Termination of Pioglitazone Therapy: Results from ACT NOW. J Clin Endocrinol Metab. 2016 May;101(5):2056-62. doi: 10.1210/jc.2015-4202. Epub 2016 Mar 16. PMID 26982008
- [Derived] Tripathy D, Cobb JE, Gall W, Adam KP, George T, Schwenke DC, Banerji M, Bray GA, Buchanan TA, Clement SC, Henry RR, Kitabchi AE, Mudaliar S, Ratner RE, Stentz FB, Reaven PD, Musi N, Ferrannini E, DeFronzo RA. A novel insulin resistance index to monitor changes in insulin sensitivity and glucose tolerance: the ACT NOW study. J Clin Endocrinol Metab. 2015 May;100(5):1855-62. doi: 10.1210/jc.2014-3824. Epub 2015 Jan 20. PMID 25603459
- [Derived] Tripathy D, Clement SC, Schwenke DC, Banerji M, Bray GA, Buchanan TA, Gastaldelli A, Henry RR, Kitabchi AE, Mudaliar S, Ratner RE, Stentz FB, Musi N, Reaven PD, DeFronzo RA. Baseline adiponectin levels do not influence the response to pioglitazone in ACT NOW. Diabetes Care. 2014 Jun;37(6):1706-11. doi: 10.2337/dc13-1745. Epub 2014 Apr 4. PMID 24705615
- [Derived] Saremi A, Schwenke DC, Buchanan TA, Hodis HN, Mack WJ, Banerji M, Bray GA, Clement SC, Henry RR, Kitabchi AE, Mudaliar S, Ratner RE, Stentz FB, Musi N, Tripathy D, DeFronzo RA, Reaven PD. Pioglitazone slows progression of atherosclerosis in prediabetes independent of changes in cardiovascular risk factors. Arterioscler Thromb Vasc Biol. 2013 Feb;33(2):393-9. doi: 10.1161/ATVBAHA.112.300346. Epub 2012 Nov 21. PMID 23175674
- [Derived] DeFronzo RA, Tripathy D, Schwenke DC, Banerji M, Bray GA, Buchanan TA, Clement SC, Henry RR, Hodis HN, Kitabchi AE, Mack WJ, Mudaliar S, Ratner RE, Williams K, Stentz FB, Musi N, Reaven PD; ACT NOW Study. Pioglitazone for diabetes prevention in impaired glucose tolerance. N Engl J Med. 2011 Mar 24;364(12):1104-15. doi: 10.1056/NEJMoa1010949. PMID 21428766
- [Derived] Defronzo RA, Banerji M, Bray GA, Buchanan TA, Clement S, Henry RR, Kitabchi AE, Mudaliar S, Musi N, Ratner R, Reaven PD, Schwenke D, Stentz FB, Tripathy D. Actos Now for the prevention of diabetes (ACT NOW) study. BMC Endocr Disord. 2009 Jul 29;9:17. doi: 10.1186/1472-6823-9-17. PMID 19640291
- See also: American Diabetes Association — http://www.diabetes.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone: Pioglitazone tablet similar to placebo tablet
  Pioglitazone: Pioglitazone tablets - 45mg/day tablet
Period: Overall Study
Arm/Group | Placebo | Pioglitazone
Started | 299 | 303
Completed | 228 | 213
Not Completed | 71 | 90

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo tablet similar to pioglitazone tablet
  Placebo: Placebo tablets similar to pioglitazone tablets
- Pioglitazone: Pioglitazone tablet similar to placebo tablet
  Pioglitazone: Pioglitazone tablets
- Total: Total of all reporting groups
Arm/Group | Placebo | Pioglitazone | Total
Number analyzed (Participants) | 299 | 303 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 269 | 271 | 540
  >=65 years | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (0.5) | 52.3 (0.5) | 52.3 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 127 | 253
  Male | 173 | 176 | 349
Region of Enrollment [Number; unit: participants]
  United States | 299 | 303 | 602

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Type 2 Diabetes
Description: Percentage of Participants with Type 2 Diabetes at 2.4 years Post-randomization
Time Frame: 2.4 years
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 299 | 303
percentage of participants | 16.1 | 5.0

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose of 2.4 Years
Description: Fasting Plasma Glucose
Time Frame: Baseline versus 2.4 years
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 299 | 303
mg/dl | -4.0 (0.09) | -10.7 (0.9)

3. Secondary Outcome: Change From Baseline in Plasma Insulin Concentration During Oral Glucose Tolerance Test
Description: Insulin secretion
Time Frame: Baseline versus 2.4 years
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 299 | 303
nmol | 35 (5) | 25 (4)

4. Secondary Outcome: Change From Baseline in Matsuda Index of Insulin Sensitivity (There Are no Minimum/Maximum Values)
Description: Insulin sensitivity The Matsuda index was calculated as 10,000/square root of (pre-meal glucose x pre-meal insulin x mean 120 min post-meal glucose x mean 120 min post-meal insulin), with higher numbers indicating better the insulin sensitivity.
Time Frame: Baseline versus 2.4 years
Measure: Mean (Standard Deviation); unit: matsuda index
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 299 | 303
matsuda index | 0.7 (0.2) | 3.6 (0.2)

5. Secondary Outcome: Change in Atherosclerosis
Description: carotid intima thickness
Time Frame: Baseline versus 2.4 years
Measure: Mean (Standard Deviation); unit: percentage of intima
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 299 | 303
percentage of intima | 1.7 (0.2) | 3.2 (0.2)

ADVERSE EVENTS:
Time Frame: 2.4 years
Arm/Group | Placebo | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 1/299 | 3/303
Other Adverse Events (participants affected / at risk) | 170/299 | 95/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=299) | Pioglitazone (N=303)
Death (General disorders) | 1 (1) | 3 (3) — One unexplained sudden death occurred in the placebo group, and three deaths occurred in the pioglitazone group (one unexplained sudden death, one death from biliary carcinoma, and one death from a carcinoid tumor).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=299) | Pioglitazone (N=303)
Myocardio infarction, heart failure, other (Cardiac disorders) | 26 (26) | 23 (23)
Other (General disorders) | 144 (144) | 72 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No